CLINICAL TRIAL: NCT05728047
Title: Evaluation of Systemic Microcirculation During the Preoperative and Early Postoperative Periods of Patients Undergoing Heart Valve Surgery
Brief Title: Evaluation of Systemic Microcirculation of Patients Undergoing Heart Valve Surgery
Status: Completed | Type: Observational
Sponsor: National Institute of Cardiology, Laranjeiras, Brazil (Other Government)
Responsible Party: Principal Investigator, Eduardo Tibirica, MD, PhD, Senior researcher, National Institute of Cardiology, Laranjeiras, Brazil
Other Study IDs: CAAE 60999822.3.0000.5272
Record Dates: First submitted 2023-01-17; First posted 2023-02-14 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Microvascular Rarefaction; Heart Valve Diseases; Extracorporeal Circulation
Keywords: microcirculation; capillary density
MeSH Terms: conditions — Microvascular Rarefaction; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Evaluation of sublingual microcirculation with side-stream dark field imaging (cytocam) — The 'Cytocam' is a hand held computer-controlled device, a third generation video-microscope, which enables real time visualisation of the in vivo microcirculation, based upon the principle of incident dark field (IDF) illumination.

SUMMARY:
The study aims to study the systemic microcirculation in adult patients hospitalized at a quaternary public hospital during the preoperative and immediate postoperative periods of heart valve surgery and correlations to their clinical and laboratory outcomes in the postoperative period.

DETAILED DESCRIPTION:
Despite the development of new endovascular procedures in recent years, cardiac surgery currently remains an important instrument in the management of patients with severe heart diseases, such as hemodynamically significant coronary obstructions and valve pathologies.

Despite the advances in the management of patients in intensive care, the postoperative period of patients undergoing cardiac surgery remains a challenge due to the intense inflammatory reaction triggered by the surgical procedure itself and exacerbated by the use of cardiopulmonary bypass (CPB), fundamental in most cardiac surgeries performed nowadays.

In this context, cardiac surgery for the treatment of valve pathologies with the use of CPB is more related to unfavorable clinical outcomes in the postoperative period in relation to coronary artery bypass grafting (CABG). It is postulated, as a causal factor, the longer CPB time in valve surgeries associated with more prominent cardiac morphological changes in these patients.

Studies carried out in recent years in patients hospitalized in intensive care that developed a severe inflammatory reaction, either due to sepsis, surgical procedure or more recently due to the Covid-19 pandemic, have shown a frequent dissociation between the hemodynamic findings measured in the ICU with the data of the patients' systemic microcirculation.

The use of portable microscopes has allowed the measurement of systemic microcirculation at the bedside in intensive care, enabling prompt assessment of aspects related to tissue perfusion, thus seeking to improve clinical outcomes in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to heart valve surgery under cardiopulmonary bypass.

Exclusion Criteria:

* Patients operated on for infective endocarditis

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to heart valve surgery under cardiopulmonary bypass.
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2022-09-10 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of systemic microcirculation | Change of microvascular density between the preoperative and up to four hours in the postoperative period.
  Number of capillaries in the sublingual microcirculation.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Cardiology, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No